CLINICAL TRIAL: NCT02436200
Title: Neuromuscular Electrical Stimulation in Patients With Intermittent Claudication
Brief Title: Neuromuscular Electrical Stimulation (NMES) in Patients With Intermittent Claudication
Acronym: IC
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Imperial College London (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 14HH1909
Record Dates: First submitted 2015-04-24; First posted 2015-05-06 (Estimated); Results first posted 2019-09-20 (Actual); Last update posted 2020-09-29 (Actual); Status verified 2020-09

CONDITIONS: Intermittent Claudication; Peripheral Vascular Disease
Keywords: Intermittent Claudication; IC; Peripheral Arterial Disease; Peripheral Vascular Disease; Peripheral Arterial Occlusive Disease
MeSH Terms: conditions — Intermittent Claudication; Peripheral Vascular Diseases; Peripheral Arterial Disease; Peripheral Arterial Occlusive Disease 1

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Intervention (Experimental): Patients receiving neuromuscular electrical stimulation.
  Interventions: Device: Neuromuscular Electrical Stimulation

INTERVENTIONS:
Device: Neuromuscular Electrical Stimulation — Revitive IX neuromuscular electrical stimulation device will be given to all participants as per protocol.

SUMMARY:
This study will assess the benefit of a neuromuscular electrical stimulation device in patients suffering from symptoms and effects of lower limb intermittent claudication.

DETAILED DESCRIPTION:
The circulation of blood around the body is dependent on effective pumping of the heart. Patients with claudication experience pain or discomfort in their legs usually during activity such as walking, which goes away at rest. Claudication is a symptom of peripheral arterial disease (PAD). If left untreated, patients can develop arterial insufficiency which can lead to various complications such as swelling, painful legs, reduced healing of injuries and the loss of limbs in extreme conditions.

PAD can be defined as a narrowing of the arteries reducing blood flow. It is most commonly due to atherosclerosis, and has associations with heart disease, stroke, and diabetes. Its incidence is estimated at 7-14% in the general population, increasing with age to about 20% in the over-seventies. It is associated with effects on mobility, skin condition and quality of life. Symptoms include pain in the legs on walking (intermittent claudication), pain at rest (particularly at night), gangrene, and limb loss. Management of PAD is based on encouraging exercise, and modification of risk factors such as smoking, high blood pressure, high cholesterol and diabetes.

In patients with PAD, exercise tolerance is often limited. Severe symptoms and disease can be treated by procedures such as balloon angioplasty, stenting or surgical bypass, but these procedures have risks. There also remains a percentage of patients who are not suitable for revascularisation, and have few options besides amputation available to them.

Some trials have shown that increasing the blood flow in the legs over time using medical devices (intermittent pneumatic compression, muscle stimulators), in addition to maximal medical and surgical therapy, can increase claudication distance, absolute walking distance, decrease rest pain, and reduce amputation rates. In our unit it has become apparent that there are an increasing number of medical devices available for circulatory support, either for use as an inpatient, out-patient, or a member of the general public. The supporting evidence for these is variable in scientific and clinical content or relevance, and requires clinical trials to evaluate further.

The device being used in this study, activates the pumping action of the leg muscles by providing neuromuscular electrical stimulation (NMES) to cause foot muscle contraction and relaxation. This squeezes blood back towards the heart, improving circulation.

The study will evaluate whether NMES using this device has the same beneficial effects in patients with intermittent claudication.

ELIGIBILITY:
Inclusion Criteria:

* All ethnic groups, male or female above the age of 18 years.
* Diagnosis of mild intermittent claudication
* Be of non-childbearing potential; OR using adequate contraception and have a negative urine pregnancy test result within 24 hours if appropriate before using the study device.
* Blood pressure currently under moderate control (< 160/100mmHg)
* No current foot ulceration

Exclusion Criteria:

* Patients meeting any of the following criteria are to be excluded:

  * Has an unstable condition (eg, psychiatric disorder, a recent history of substance abuse) or otherwise thought to be unreliable or incapable of complying with the study protocol.
  * Has diabetes
  * Ankle Brachial Pressure Index > 0.9
  * Has any metal implants
  * Pregnant
  * Has a cardiac pacemaker or defibrillator device
  * Has recent lower limb injury or lower back pain
  * Has current foot ulceration or other skin ulcers
  * Has foot deformities
  * Has any disorder that, in the opinion of the Investigator, might interfere with the conduct of the study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 21 (Actual)
Dates: Start 2014-12 (Actual); Primary Completion 2015-10 (Actual); Study Completion 2015-10 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Alun H Davies, BA BMChB MA, Study Chair — Imperial College London
Locations (1):
- Imperial College London - Charing Cross Hospital, London, Hammersmith, United Kingdom

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Babber A, Ravikumar R, Onida S, Lane TRA, Davies AH. Effect of footplate neuromuscular electrical stimulation on functional and quality-of-life parameters in patients with peripheral artery disease: pilot, and subsequent randomized clinical trial. Br J Surg. 2020 Mar;107(4):355-363. doi: 10.1002/bjs.11398. Epub 2020 Jan 7. PMID 31912491

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Intervention
Started | 21
Completed | 20
Not Completed | 1
Not completed — Significant outlier | 1

BASELINE CHARACTERISTICS:
Arm/Group | Intervention
Number analyzed (Participants) | 20
Age, Continuous [Mean (Standard Deviation); unit: years] | 70 (11.7)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 4
  Male | 16
Region of Enrollment [Number; unit: participants]
  United Kingdom | 20
Body Mass Index - BMI [Mean (Standard Deviation); unit: kg/m^2] | 27.4 (4.5)
Ankle Brachial Pressure Index - ABPI (Right) [Mean (Standard Deviation); unit: Ratio] — The ankle-brachial index test is a quick, noninvasive way to check for peripheral artery disease (PAD). The ankle-brachial index test compares the blood pressure measured at the ankle with the blood pressure measured at the arm.
  Ratio | 0.71 (0.17)
Ankle Brachial Pressure Index - ABPI (Left) [Mean (Standard Deviation); unit: Ratio] | 0.69 (0.17)
Initial Claudication Distance - ICD (m) [Median (Inter-Quartile Range); unit: m] | 37.7 [29 to 64.45]
Maximum Claudication Distance - MCD (m) [Median (Inter-Quartile Range); unit: m] | 89.3 [57.8 to 138.1]

OUTCOME MEASURES:

1. Primary Outcome: Change From Baseline in Initial Walking Distance
Description: Initial walking distance measured by treadmill For the initial claudication distance measurement, a fixed load treadmill test will be carried out at 3.5 km/h with a 10% gradient. The initial claudication distance (ICD) is the distance walked until the onset of pain.
Time Frame: Baseline, 6 weeks
Measure: Median (Inter-Quartile Range); unit: metres
Arm/Group | Intervention
Number analyzed (Participants) | 20
metres | 64.3 [48 to 132]

2. Primary Outcome: Absolute Walking Distance Measured by Treadmill
Description: For the absolute claudication distance measurement, a fixed load treadmill test will be carried out at 3.5 km/h with a 10% gradient. The absolute claudication distance (ACD) is the distance walked before the participant is forced to stop due to typical pain.
Time Frame: Change in baseline treadmill walking distance at 6 weeks
Measure: Median (Inter-Quartile Range); unit: m
Arm/Group | Intervention
Number analyzed (Participants) | 20
m | 130 [85.9 to 281.2]

3. Secondary Outcome: Femoral Haemodynamics Measured by Femoral Artery Duplex Ultrasonography
Description: Ultrasound assessment of blood flow dynamics in the femoral artery will be obtained at rest, and if randomised to the intervention group, whilst using the device.
Time Frame: Change in baseline femoral haemodynamics at 6 weeks
Reporting Status: Not Posted

4. Secondary Outcome: Laser Doppler Flow Measured by Optical Laser
Description: Optical laser flowmetry probes will be used to assess the superficial skin circulation and temperature.
Time Frame: Change in baseline flowmetry at 6 weeks
Reporting Status: Not Posted

5. Secondary Outcome: Symptomatic Scores by Questionnaire
Description: Validated questionnaires including the Edinburgh Claudication Questionnaire and Intermittent Claudication Questionnaire will be obtained at baseline and week 6.
Time Frame: Change in baseline questionnaire scores at 6 weeks
Reporting Status: Not Posted

6. Secondary Outcome: Quality of Life Scores Measured by Questionnaire
Description: Validated questionnaires including the Euro-Quol 5D and Short Form 36 will be measured at baseline and 6 weeks.
Time Frame: Change in baseline quality of life at 6 weeks
Reporting Status: Not Posted

7. Secondary Outcome: Urine Metabolic Profile
Description: A urine sample will be collected at baseline and at 6 weeks. Mass spectroscopy and nuclear magnetic resonance spectroscopy analysis will be carried out.
Time Frame: Change of profile at baseline and at 6 weeks
Reporting Status: Not Posted

8. Secondary Outcome: Serum Metabolic Profile
Description: A serum sample will be collected at baseline and at 6 weeks. Mass spectroscopy and nuclear magnetic resonance spectroscopy analysis will be carried out.
Time Frame: Change of profile at baseline and 6 weeks
Reporting Status: Not Posted

ADVERSE EVENTS:
Time Frame: 6 weeks - duration of study
Arm/Group | Intervention
All-Cause Mortality (participants affected / at risk) | 0/20
Serious Adverse Events (participants affected / at risk) | 0/20
Other Adverse Events (participants affected / at risk) | 0/20

LIMITATIONS AND CAVEATS:
Small scale pilot study.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes